CLINICAL TRIAL: NCT02354118
Title: Maintaining Patency in Implanted Port Catheters With Saline Only Flushes
Brief Title: Maintaining Patency in Implanted Port Catheters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Principal Investigator, Rachel Baker, Nurse Researcher, TriHealth Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12135-12-079
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Results first posted 2022-09-14 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-09

CONDITIONS: Obstruction; Catheter, Infusion Catheter (Vascular); Catheter; Complications (Indwelling Catheter)
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Active Comparator): Heparinized saline catheter flush - The control group will have their port catheters flushed with 20mL saline + 5mL heparin 100 units/mL; q 3 months
  Interventions: Other: Heparinized saline catheter flush
- Intervention Group (Experimental): Saline-only catheter flush - The intervention group will have their port catheters flushed with saline only.
  Interventions: Other: Saline-only catheter flush

INTERVENTIONS:
Other: Heparinized saline catheter flush — The control group will have their port catheters flushed with 20mL saline + 5mL heparin 100 units/mL; q 3 months
  Arms: Control Group
Other: Saline-only catheter flush — The intervention group will have their port catheters flushed with saline only.
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to determine the safest and most effective flushing solution for maintaining patency (unobstructed flow) in implanted port catheters. The complication rate in patients whose ports are flushed with saline only will be compared to the complication rate in patients whose ports are flushed with a combination of saline and heparinized saline.

DETAILED DESCRIPTION:
The purpose of this study is to determine the safest and most effective flushing solution for maintaining patency (unobstructed flow) in implanted port catheters. The complication rate in patients whose ports are flushed with saline only will be compared to the complication rate in patients whose ports are flushed with a combination of saline and heparinized saline. These complications include partial or complete obstruction, infection of the central line, and/or the onset of heparin induced thrombocytopenia.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and understand English
* Has an implanted port in place less than one (1) year
* Evidence of a patent (unobstructed) port catheter prior to enrollment in the study
* Is receiving active treatment (i.e., receiving a therapeutic drug through the implanted port)
* Current treatment protocol projected to continue for a minimum of three (3) months
* Anticipates receiving care at the identified centers for 12 months following enrollment in the study
* Does not receive care of implanted port at any other facility

Exclusion Criteria:

* Has documented heparin platelet antibody (i.e., could not be randomized to either group) or other allergy to heparin
* Receiving therapeutic dose of an anticoagulant (e.g.,warfarin, heparin, enoxaparin)
* Does not have a BioFlo port (heparinized port)
* Does not meet one or more of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2021-12-11 (Actual); Study Completion 2021-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Pelgen, BSN, RN, OCN, Principal Investigator — TriHealth Cancer Institute
Locations (8):
- United States (8):
  - UC Health Barrett Infusion Center, Cincinnati, Ohio
  - TriHealth Cancer Institute Good Samaritan Infusion Center at GSH, Cincinnati, Ohio
  - Ambulatory Treatment Center at Bethesda North TriHealth Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute Good Samaritan Infusion Center, Medicenter, Cincinnati, Ohio
  - TriHealth Cancer Institute Good Samaritan Infusion Center, Cheviot, Cincinnati, Ohio
  - TriHealth Cancer Institute Good Samaritan Infusion Center, Anderson, Cincinnati, Ohio
  - TriHealth Cancer Institute Good Samaritan Infusion Center Butler County, Hamilton, Ohio
  - McCullough Hyde Memorial Hospital Infusion Center, Oxford, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Intervention Group
Started | 222 | 214
Completed | 222 | 214
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group | Total
Number analyzed (Participants) | 222 | 214 | 436
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.14 (12.32) | 59.30 (11.61) | 59.22 (11.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 153 | 143 | 296
  Male | 69 | 71 | 140
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 222 | 214 | 436

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Complete Occlusion Within 1 Year
Description: Number of participants who had a first complete occlusion (Blockage) within 1 year
Time Frame: baseline to 1 year
Population: NOTE: 1 participant had BOTH a partial occlusion and a complete occlusion. Therefore, when adding information from Outcome Measures 1 and 2 to determine the total number of participants with either complete or partial occlusions in the "Control Group" is correct as 43 (i.e., (5+39 = 44) - 1 participant in both groups = 43 distinct participants)
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 222 | 214
Participants | 5 | 4

2. Primary Outcome: Number of Participants With First Partial Occlusion Within 1 Year
Description: Number of Participants with First Partial Occlusion (Blockage) within 1 year
Time Frame: baseline to 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 222 | 214
Participants | 39 | 55

3. Primary Outcome: Number of Participants With First Cathflo Administration for Occlusion (Blockage) Within 1 Year
Description: Number of Participants with First Cathflo administration for Occlusion (Blockage) within 1 year
Time Frame: baseline to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 222 | 214
Participants | 39 | 55

4. Secondary Outcome: Number of Participants With First Complete or Partial Occlusion Within 1 Year
Description: Number of Participants with either a First Complete or Partial Occlusion (Blockage) within 1 year
Time Frame: baseline to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 222 | 214
Participants | 43 | 59

5. Secondary Outcome: Number of Participants With HIT Within 1 Year
Description: Heparin Induced Thrombocytopenia (HIT) as measured by a positive HIT antibody test, or any other heparin allergy, will be recorded.
Time Frame: baseline to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 222 | 214
Participants | 0 | 0
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Non-Inferiority — 10% non-inferiority margin; p = 1.0, Chi-squared

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Control Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 42/222 | 27/214
Serious Adverse Events (participants affected / at risk) | 0/222 | 0/214
Other Adverse Events (participants affected / at risk) | 0/222 | 0/214

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT02354118/Prot_SAP_000.pdf